CLINICAL TRIAL: NCT04579510
Title: Immunogenicity of Novel Monovalent Oral Poliovirus Vaccine Type 2 (nOPV2) With and Without Bivalent OPV
Brief Title: Immunogenicity nOPV2 With and Without bOPV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20060
Record Dates: First submitted 2020-09-22; First posted 2020-10-08 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Poliomyelitis
Keywords: oral poliovirus vaccine; immunization; antibodies; poliovirus vaccines
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- nOPV2 only (Active Comparator): Participants in this arm will receive nOPV2 at 6, 10, and 14 weeks of age
  Interventions: Biological: Novel monovalent oral poliovirus vaccine type 2 (nOPV2)
- nOPV2 and bOPV (Active Comparator): Participants in this arm will receive both nOPV2 and bOPV at 6, 10, and 14 weeks of age
  Interventions: Biological: Novel monovalent oral poliovirus vaccine type 2 (nOPV2); Biological: Bivalent oral poliovirus vaccine (bOPV)
- bOPV only (Active Comparator): Participants in this arm will receive bOPV at 6, 10, and 14 weeks of age
  Interventions: Biological: Bivalent oral poliovirus vaccine (bOPV)

INTERVENTIONS:
Biological: Novel monovalent oral poliovirus vaccine type 2 (nOPV2) — nOPV2 candidate 1 (S2/cre5/S15domV/rec1/hifi3) is a live-attenuated serotype-2 poliovirus that was derived from a modified Sabin type-2 infectious cDNA clone and propagated in Vero cells. To improve genetic stability, nucleotide sequence modifications were made in the major determinant for attenuation in the Sabin 5'-untranslated region. Additionally, two modifications in the polymerase 3D were made to further improve stability of the attenuation, and a key replication element from the 2C coding region was relocated to the 5'-untranslated region to inhibit recombination.
  Arms: nOPV2 and bOPV; nOPV2 only
Biological: Bivalent oral poliovirus vaccine (bOPV) — The live types 1 & 3 oral polio vaccine (bOPV) is a bivalent vaccine containing suspension of types 1 & 3 attenuated Polio viruses (Sabin strains).
  Arms: bOPV only; nOPV2 and bOPV

SUMMARY:
This is an open-label randomized clinical trial that will compare immune responses among infants who receive either novel monovalent oral poliovirus vaccine type 2 (nOPV2) alone, bivalent oral poliovirus vaccine (bOPV) alone, or co-administered nOPV2 and bOPV.

DETAILED DESCRIPTION:
It is expected that nOPV2 would replace mOPV2 for responding to type 2 outbreaks. Outbreak response for cVDPV2 also offers the opportunity to close immunity gaps to polioviruses types 1 and 3. Furthermore, GPEI might have to respond to two poliovirus outbreaks in the same geography. For either scenario, it would be important to get data on the immunogenicity of co-administered nOPV2 and bOPV, compared to either vaccine given alone.

This clinical trial assesses and compares the immunogenicity of nOPV2 given with or without bOPV. Healthy infants 6 weeks of age will be enrolled in Dhaka, Bangladesh, and randomized to one of three study arms â " Arm A: nOPV2 only, Arm B: nOPV2 and bOPV, or Arm C: bOPV only. Infants will be followed-up until 18 weeks of age through clinic and household visits. Blood specimens will be collected to test for immunological response. Stool specimens will be collected from infant vaccine recipients and one sibling household contact each to assess viral recombinants and nOPV2 household transmission.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 6 weeks of age (range: 42-48 days).
* Parents that consent for participation in the full length of the study.
* Parents that can understand and comply with planned study procedures.
* Infant has at least one sibling aged <10 years living in the same household that is eligible for participation in the study.

Exclusion Criteria:

* Parents and infants who are unable to participate in the full length of the study (e.g., plan to move away from the study area during the study period).
* A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member.
* A diagnosis or suspicion of bleeding disorder that would contraindicate administration of bOPV or nOPV2 or collection of blood by venipuncture.
* Acute diarrhoea, infection or illness at the time of enrolment (6 weeks of age) that would require infant's admission to a hospital.
* Acute vomiting and intolerance to liquids within 24 hours before the enrolment visit (6 weeks of age).
* Evidence of a chronic medical condition identified by a study medical officer during physical exam.
* Receipt of any polio vaccine (OPV or IPV) before enrolment based upon documentation or parental recall.
* Known allergy/sensitivity or reaction to polio vaccine, or its contents.
* Infants from multiple births. Infants from multiple births will be excluded because the infant(s) who is/are not enrolled would likely receive OPV through routine immunization and transmit vaccine poliovirus to the enrolled infant. Even if all births from a multiple birth could be enrolled in the study, we will exclude multiple births as discontinuation of one may lead to discontinuation of multiple participants.
* Infants from premature births (<37 weeks of gestation).

Ages: 42 Days to 48 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 795 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Vaccine response | Measured four weeks after administration of study vaccine(s).
  Dichotomous (yes/no) variable defined as participants who are either seronegative (<1:8 titers) at baseline who become seropositive (≥1:8) after vaccination (seroconversion) or participants who demonstrate a four-fold rise in titers after vaccination between two specimens, e.g. a change from 1:8 to 1:32, after adjusting for expected decay in maternal antibodies. Antibody titers at 6 weeks of age will be the starting point for the expected decline in maternal antibodies, assuming at half-life of 28 days.

SECONDARY OUTCOMES:
Reciprocal antibody titers | Measured four weeks after administration of study vaccine(s).
  Variable of the observed reciprocal antibody titer results.
Household transmission of nOPV2 | 1, 2, and 4 weeks after first vaccination with nOPV2
  Detection of type 2 OPV in stool of household contact
Viral recombinants | 2 and 4 weeks after first vaccination with study vaccine(s)
  Detection and characterization of viral recombinants

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Wilkinson, PhD, Principal Investigator — Centers for Disease Control and Prevention; Khalequ Zaman, MBBS, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddr,B Study Clinics, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Aggregated data will be added to the registration with publication. In accordance with the protocol, icddr,b investigators will have access to participant data with identifiers. External investigators will have access to deidentified participant data. Deidentified data may be shared with national and international vaccine manufacturers and regulatory authorities upon request.

REFERENCES:
- [Derived] Wilkinson AL, Zaman K, Hoque M, Estivariz CF, Burns CC, Konopka-Anstadt JL, Mainou BA, Kovacs SD, An Q, Lickness JS, Yunus M, Snider CJ, Zhang Y, Coffee E, Abid T, Wassilak SGF, Pallansch MA, Oberste MS, Vertefeuille JF, Anand A. Immunogenicity of novel oral poliovirus vaccine type 2 administered concomitantly with bivalent oral poliovirus vaccine: an open-label, non-inferiority, randomised, controlled trial. Lancet Infect Dis. 2023 Sep;23(9):1062-1071. doi: 10.1016/S1473-3099(23)00139-1. Epub 2023 May 10. PMID 37178706

DOCUMENTS (1):
  • Study Protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT04579510/Prot_000.pdf